CLINICAL TRIAL: NCT06581640
Title: A Clinical Study of the Safety and Efficacy of Chimeric Antigen Receptor-modified T Cells Targeting BCMA for the Treatment of Relapsed/Refractory Multiple Myeloma
Brief Title: Chimeric Antigen Receptor Modified T Cells Targeting BCMA for the Treatment of Relapsed/Refractory Multiple Myeloma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Principal Investigator, Bing, Xu, Principal Investigator, The First Affiliated Hospital of Xiamen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMDYYYXYK-11
Record Dates: First submitted 2024-08-30; First posted 2024-09-03 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma; Relapsed/Refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T (Experimental)
  Interventions: Biological: CAR-T treatment

INTERVENTIONS:
Biological: CAR-T treatment — Peripheral blood lymphocyte collection, PBMC separation, BCMA CAR-T cell preparation/storage, lymphodepletion chemotherapy pretreatment for the subject, and BCMA CAR-T cell infusion.

SUMMARY:
To evaluate the safety and tolerability of chimeric antigen receptor gene-modified T cells targeting BCMA for the treatment of relapsed/refractory multiple myeloma

DETAILED DESCRIPTION:
Subjects who meet the eligibility criteria, PBMC will be collected by blood cell separator and 50 mL of plasma will be collected for preparation of CAR-T and frozen storage of CAR-T preparations; patients will be treated with autologous BCMA CAR-T transfusion and followed up for a period of 3 years, with specific efficacy judgments referring to the IMWG Clinical Efficacy Evaluation Criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, no gender restrictions;
2. Diagnosed with refractory/relapsed multiple myeloma through physical examination, pathological examination, laboratory tests, and imaging studies;
3. Flow cytometry or histology confirms positive BCMA expression in myeloma cells;
4. As judged by the investigator, the expected survival time is >3 months;
5. ECOG performance status score ≤2, KPS >60%;
6. The patient has good liver, kidney, heart, and lung function: ALT and AST ≤2.5×ULN, those with liver involvement can be relaxed to ≤5×ULN; serum total bilirubin <34 μmol/L; creatinine clearance rate >30 mL/min; heart ejection fraction (EF) ≥40%, no pericardial effusion and significant arrhythmia; indoor SpO2 ≥92%;
7. Peripheral blood lymphocyte absolute count ALC ≥0.5 ×10^9/L, PLT >30×10^9/L, Hb >80 g/L and has a single collection venous access, and there are no other contraindications for hematopoietic cell separation;
8. Those with fertility must agree to use highly effective contraceptive methods;
9. The subject or their legal guardian can understand and is willing to sign a written informed consent form voluntarily.

Exclusion Criteria:

1. Pregnant or nursing women, as well as women planning to become pregnant within the next six months;
2. Positive virology tests for hepatitis B, hepatitis C, HIV, syphilis, or cytomegalovirus;
3. History of other tumors (except for those with skin or cervical in situ cancers that have been cured by radical treatment and show no evidence of disease activity);
4. Previously received treatment targeting BCMA;
5. Underwent autologous hematopoietic stem cell transplantation within the last 6 weeks;
6. Presence of uncontrolled active bacterial or fungal infection;
7. Allergic to research-related drugs or cell components;
8. Presence of active autoimmune diseases;
9. Currently have unstable or active ulcers or gastrointestinal bleeding;
10. Unable to cooperate with treatment and efficacy evaluation due to mental or psychological disorders;
11. Received other experimental drug treatments within the last 3 months;
12. The researcher believes that for other reasons, the individual is not suitable for the clinical trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-09-24 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate (CR) | Up to 36 months
  Negative serum and urine immunofixation electrophoresis, disappearance of soft tissue plasmacytoma, and less than 5% plasma cells in the bone marrow. For patients who rely solely on serum FLC levels as a measurable lesion, in addition to meeting the above CR criteria, it is also required that the ratio of serum FLC is restored to normal in two consecutive evaluations.

SECONDARY OUTCOMES:
Adverse events (AE) | Up to 36 months
  Any adverse and unexpected signs, symptoms, or diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Xu, Principal Investigator — The First Aiffiliated hosptical of xiamen University
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China